CLINICAL TRIAL: NCT06839573
Title: Effectiveness of Immersive Virtual Reality to Improve Learning Outcomes in Nursing Degree Students: A Randomized Clinical Trial
Brief Title: Effectiveness of Immersive Virtual Reality in Nursing Students' Learning
Acronym: UBUJIRV25
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: University of Barcelona (Other); Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Isabel Almodóvar Fernández, Principal Investigator, Universitat Jaume I
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: UB-UJI-RV25
Record Dates: First submitted 2025-01-25; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Informed Consent
Keywords: Virtual reality; nursing students; Learning Outcomes; Inmersive virtual reality

STUDY DESIGN:
Intervention Model Description: Open, single-center randomized clinical trial involving fourth-year nursing degree students at a public university. Participants will be assigned based on their usual teaching groups (ratio of 6-8 students per instructor) and, according to randomization, will receive a 1:1 assignment to either the control group (classroom-based simulation teaching) or the experimental group (classroom-based simulation teaching combined with VR headset teaching). The CONSORT checklist will be followed to report the study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RV INTERVENTION (Experimental): Experience with virtual reality glasses
  Interventions: Other: Experience with virtual reality glasses
- NON RV CONTROL (No Intervention): Group Control

INTERVENTIONS:
Other: Experience with virtual reality glasses — If the group belongs to GE (teaching with in-person simulation in the classroom and teaching with VR headsets), they will also receive the two training sessions described for GC:
  30 minutes of individual training through VR (headsets and controllers to perform actions while receiving immediate feedback through VR) before the in-person simulation.
  Other Names: Formative intervention
  Arms: RV INTERVENTION

SUMMARY:
Teaching using VR for basic cardiopulmonary resuscitation and patient examination (experimental group) will not result in differences in knowledge and skill acquisition compared to traditional classroom-based simulation teaching (control group), but it will lead to greater satisfaction and self-confidence. Open, single-center randomized clinical trial involving fourth-year nursing degree students at a public university. Participants will be assigned based on their usual teaching groups (ratio of 6-8 students per instructor) and, according to randomization, will receive a 1:1 assignment to either the control group (classroom-based simulation teaching) or the experimental group (classroom-based simulation teaching combined with VR headset teaching). The CONSORT checklist will be followed to report the study.

ELIGIBILITY:
Inclusion Criteria:

- having completed the scheduled in-person simulation in previous years of the degree .

Exclusion Criteria:

-the student does not sign the informed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-03-05 (Estimated); Primary Completion 2025-03-05 (Estimated); Study Completion 2025-05-08 (Estimated)

PRIMARY OUTCOMES:
Compare the satisfaction | Five months
  To compare the satisfaction acquired by students when performing basic cardiopulmonary resuscitation and patient examination between both teaching groups (experimental group - EG: VR plus in-person simulation, control group - CG: in-person simulation). We will mesure this with Satisfaction and Self-Confidence in Learning Scale (SCLS-Sp) (Farrés-Tarafa et al., 2021) .
Compare the self-confidence | Five months
  To compare the self-confidence acquired by students when performing basic cardiopulmonary resuscitation and patient examination between both teaching groups (experimental group - EG: VR plus in-person simulation, control group - CG: in-person simulation). We will mesure this with Satisfaction and Self-Confidence in Learning Scale (SCLS-Sp) (Farrés-Tarafa et al., 2021) .

SECONDARY OUTCOMES:
To compare the acquisition of knowledge in each teaching group. | Five months
  We will use the Knowledge and Skills Checklist to perform basic CPR to measure. Adapted from European Resuscitation Council Guidelines (Perkins et al., 2021), with official translation into Spanish from the Spanish CPR Council and validated in the Boada study (Boada et al., 2015). CPR instructor faculty who does not participate in simulation-based teaching will evaluate the performance in situ of the group during the face-to-face simulation scenario.
To compare the acquisition of skills in each teaching group. | Five months
  We will use the Knowledge and Skills Checklist to perform basic CPR to measure. Adapted from European Resuscitation Council Guidelines (Perkins et al., 2021), with official translation into Spanish from the Spanish CPR Council and validated in the Boada study (Boada et al., 2015). CPR instructor faculty who does not participate in simulation-based teaching will evaluate the performance in situ of the group during the face-to-face simulation scenario.
To evaluate students' tolerance to VR headset technology. | Five months
  To measure this objective, we will use the Student Tolerance Scale for Teaching with VR Glasses used by Martí-Hereu (Martí-Hereu et al., 2024). Evaluate the presence of effects collaterals of the use of VR glasses with six items (nausea, dizziness drowsiness, headache, tranquility, well-being) using a scale Likert (never, rarely, sometimes, most of the time). It will be administered to the students individually at the end of teaching with the VR glasses in both teaching groups (GC after simulation in person; GE before the face-to-face simulation).
To assess the usability of VR headsets by students. | Five months
  USE questionnaire to assess the usefulness, satisfaction and ease of use of a digital technology, developed by Gao (Gao et al., 2018) and adapted to the use of immersive VR glasses with health sciences professionals by Peek (Peek et al., 2023). Scale to assess affinity with technology (ATI scale), validated to our cultural context (Franke et al., 2019).
To analyze the costs of traditional teaching with in-person simulation compared to teaching with VR. | Five months
  With all the results we will be able to analyze the cost-benefit of this new technology.

IPD SHARING:
Plan to Share IPD: Yes
The study is multicenter, so it is already planned to be shared with other researchers.
Supporting Information: CSR